CLINICAL TRIAL: NCT01542827
Title: Danish: Integreret Motion på Arbejdspladsen (IRMA) English: Implementation of Exercise at the Workplace
Brief Title: Acute Effect of Topical Menthol on Neck Pain
Acronym: IRMA04
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources to perform the study
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Marquette University (Other); Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Principal Investigator, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRMA04
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Disorders
Keywords: neck pain; menthol
MeSH Terms: conditions — Musculoskeletal Diseases; Neck Pain | interventions — Analgesics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Topical gel containing a menthol scent, but no active menthol
  Interventions: Other: Placebo
- Biofreeze (Experimental): Biofreeze topical gel containing 3.5% menthol
  Interventions: Other: Biofreeze

INTERVENTIONS:
Other: Biofreeze — The gel will be applied at 2.5 ml per 500 cm2 to the upper trapezius and neck muscles by a gloved technician
  Other Names: Topical analgesic
  Arms: Biofreeze
Other: Placebo — The gel will be applied at 2.5 ml per 500 cm2 to the upper trapezius and neck muscles by a gloved technician
  Arms: Placebo

SUMMARY:
Topical menthol gels are classified 'topical analgesics' and are used to relieve aching and tenderness of muscles and joints. However, double-blind randomized controlled trials are lacking. Here the investigators examine - in a double-blind randomized controlled cross-over trial - the acute effect of topical menthol (Biofreeze) and placebo (gel with a menthol scent) on neck pain.

ELIGIBILITY:
Inclusion Criteria:

* more than 30 days with neck pain during the last year
* frequent pain or discomfort, defined as at least 3 days per week
* pain intensity at least 4 on a scale of 0-10
* working at least 30 hours per week

Exclusion Criteria:

* blood pressure above 160/100 mmHg
* pregnancy
* life-threatening disease

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity (scale 0-10) | before and 20 min after application
  the participant rates pain intensity on a scale from 0-10 immediately before, and 0, 10, 20, 40 and 60 minutes after application of the gel. The primary efficacy endpoint is at 20 min

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | before and 20 min after application
  pressure pain threshold of the upper trapezius muscle is measured by a handheld algometer immediately before, and 0, 10, 20, 40 and 60 minutes after application of the gel.

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — Professor
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- See also: Company website — http://arbejdsmiljoforskning.dk